CLINICAL TRIAL: NCT01550614
Title: A Randomized, Controlled, Parallel Group, Multicenter Phase 3 Study to Evaluate the Efficacy and Safety of Ad5FGF-4 Using SPECT Myocardial Perfusion Imaging in Patients With Stable Angina Pectoris
Brief Title: Efficacy and Safety of Ad5FGF-4 for Myocardial Ischemia in Patients With Stable Angina Due to Coronary Artery Disease
Acronym: ASPIRE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Cardium Therapeutics (Industry)
Collaborators: Advanced Biosciences Research (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT-3-002
Record Dates: First submitted 2012-02-29; First posted 2012-03-12 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Angina, Stable
Keywords: Angina Pectoris; Myocardial Ischemia; Chest Pain; Coronary Artery Disease; Heart Diseases; Cardiovascular Diseases; Myocardial Perfusion; Reversible Perfusion Defect Size; SPECT-MIBI; Anti-Anginal Medication; Quality of Life
MeSH Terms: conditions — Angina, Stable; Angina Pectoris; Myocardial Ischemia; Chest Pain; Coronary Artery Disease; Heart Diseases; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: Ad5FGF-4 (Experimental): Adenovirus serotype-5 mediated human fibroblast growth factor-4 gene transfer and standard of care angina medication
  Interventions: Genetic: Alferminogene tadenovec
- Arm B (No Intervention): Standard of care angina medication

INTERVENTIONS:
Genetic: Alferminogene tadenovec — One-time intracoronary infusion of Ad5FGF-4 (6x10e9 viral particles in buffer)
  Other Names: Generx; Cardionovo (Russian Trade Name)
  Arms: Arm A: Ad5FGF-4

SUMMARY:
The purpose of this study is to determine whether a single intracoronary infusion of Ad5FGF-4, delivered during induced transient ischemia, is effective in improving myocardial perfusion, angina functional class, patient symptoms, and quality of life. Short-term (8 weeks) and long-term (12 month) safety of Ad5FGF-4 will also be evaluated. The primary endpoint is change in adenosine triphosphate (ATP) stress SPECT reperfusion defect size.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18-75 years of age, inclusive
* Postmenopausal female patients, women of childbearing potential and men willing to use an effective contraception method while on the study treatment and/or who agree not to become pregnant or make their partner pregnant throughout the study and during one year after administration of the study drug
* Female subjects of childbearing potential who have a negative urine pregnancy test, and are willing to use an acceptable form of birth control during the study
* Diagnostic coronary angiogram in the past confirming the presence of coronary artery disease. Patients with extensive disease, or high risk for intervention, or who don't want the higher risk angioplasty or surgery, or have had angioplasty with recurrent angina and vessels are not ideal for angioplasty are ideal candidates
* Stable angina pectoris being treated with chronic anti-anginal medication(s) at a stable dose for 2 weeks prior to randomization
* Left ventricular ejection fraction (LVEF) of ≥30%. If the LVEF is <30% the patient can be enrolled if there is no recent or current congestive heart failure present
* Evidence of stress induced myocardial ischemia by ATP technetium-99m sestamibi SPECT, defined as a reversible perfusion defect size of ≥9%
* Willing and able to comply with the study requirements
* Provided written informed consent

Exclusion Criteria:

* Female patients who are pregnant, lactating (breast milk feeding), or planning a pregnancy during the course of the study and one year after administration of the study drug. Women of child bearing potential who are not using an acceptable method of birth control. Women of child bearing potential with a positive urine pregnancy test within 24 hours prior to the start of investigational product
* Patients with unstable angina for whom an immediate revascularization procedure is indicated
* Patients for whom a cardiac revascularization procedure is planned in the next 3 months
* Myocardial infarction within the 3 months prior to the Screening visit
* Congestive heart failure NYHA Class IV
* Myocarditis or restrictive pericarditis
* Left main coronary stenosis ≥70% (unless the patient has a patent graft or collateral vessels supplying the left coronary circulation) or proximal stenoses ≥70% in all major coronary conduit vessels (coronary arteries and bypass grafts)
* A single patent coronary conduit (for example, totally occluded RCA and LCx with no bypass grafts. Patient will not tolerate balloon occlusion of the LAD for infusion)
* Clinically significant aortic or mitral valvular heart disease.
* Life threatening coronary ostial stenosis that precludes adequate catheter engagement in any target vessel, unless the vessel can be accessed via a patent bypass graft
* Coronary artery to venous communications, which bypass the coronary capillary bed
* Untreated life-threatening ventricular arrhythmias
* Uncontrolled arterial hypertension with systolic blood pressure >180 mm Hg and diastolic pressure >100 mm Hg
* CABG surgery within the past 6 months, unless those grafts are now occluded
* Percutaneous transluminal coronary angioplasty (PTCA) within the past 3 months, unless the stented/dilated vessel(s) are now occluded
* Enhanced external counterpulsation (EECP) within 3 months prior to the start of screening evaluations
* Transmyocardial or percutaneous myocardial laser revascularization within the previous year
* Prior treatment with any cardiovascular gene therapy
* Patients who received an investigational drug or biologic within 30 days of screening or are currently participating in an investigational drug, biologic or device trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2012-03; Primary Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change in reversible perfusion defect size (RPDS) as measured by adenosine triphosphate (ATP) single-photon emission computed tomography with technetium-99m sestamibi (SPECT) | Baseline and Week 8

SECONDARY OUTCOMES:
Change in angina frequency and nitroglycerin use | Baseline and Week 8
Change in quality of life using the Seattle Angina Questionnaire | Baseline and Week 8
Change in patient functional class using CCS anginal classification | Baseline and Week 8
Safety of Ad5FGF-4 as assessed by adverse events and clinical laboratory testing | Through Week 8
Long-term safety of Ad5FGF-4 as assessed by serious adverse events | Through Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Gabor Rubanyi, Study Director — Cardium Therapeutics
Locations (1):
- Municipal Hospital #15, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Henry TD, Grines CL, Watkins MW, Dib N, Barbeau G, Moreadith R, Andrasfay T, Engler RL. Effects of Ad5FGF-4 in patients with angina: an analysis of pooled data from the AGENT-3 and AGENT-4 trials. J Am Coll Cardiol. 2007 Sep 11;50(11):1038-46. doi: 10.1016/j.jacc.2007.06.010. Epub 2007 Aug 24. PMID 17825712
- [Background] Grines CL, Watkins MW, Mahmarian JJ, Iskandrian AE, Rade JJ, Marrott P, Pratt C, Kleiman N; Angiogene GENe Therapy (AGENT-2) Study Group. A randomized, double-blind, placebo-controlled trial of Ad5FGF-4 gene therapy and its effect on myocardial perfusion in patients with stable angina. J Am Coll Cardiol. 2003 Oct 15;42(8):1339-47. doi: 10.1016/s0735-1097(03)00988-4. PMID 14563572
- [Background] Grines CL, Watkins MW, Helmer G, Penny W, Brinker J, Marmur JD, West A, Rade JJ, Marrott P, Hammond HK, Engler RL. Angiogenic Gene Therapy (AGENT) trial in patients with stable angina pectoris. Circulation. 2002 Mar 19;105(11):1291-7. doi: 10.1161/hc1102.105595. PMID 11901038
- [Derived] Kaski JC, Consuegra-Sanchez L. Evaluation of ASPIRE trial: a Phase III pivotal registration trial, using intracoronary administration of Generx (Ad5FGF4) to treat patients with recurrent angina pectoris. Expert Opin Biol Ther. 2013 Dec;13(12):1749-53. doi: 10.1517/14712598.2013.827656. Epub 2013 Aug 19. PMID 23957658